CLINICAL TRIAL: NCT00357097
Title: A Multicenter 3:1-randomized Placebo-controlled Double-blind Phase IIIb Study on the Effects of Ropinirole on Mood/(Subclinical) Depression in the Therapy of Patients With Moderate to Severe Idiopathic RLS in Germany
Brief Title: The Effects Of Ropinirole On Mood Or Mild Depression In Patients With Moderate To Severe Restless Legs Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RRL106721
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Results first posted 2009-09-16 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2011-05

CONDITIONS: Restless Legs Syndrome; Moderate to Severe Idiopathic Restless Legs Syndrome (RLS)
Keywords: randomised; ropinirole; depression; RLS; placebo; mood; double-blind; restless legs syndrome; germany
MeSH Terms: conditions — Restless Legs Syndrome; Depression | interventions — ropinirole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropinirole

SUMMARY:
Ropinirole has shown to improve mood in depressed patients as well as to improve the symptoms of Restless Legs Syndrome. Up to 40% of RLS patients suffer from mild depression, therefore it would be important for decisions no therapy to know whether a drug could improve both depressive and RLS symptoms.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of idiopathic Restless Legs Syndrome, confirmed by a score of at least 11 on the RLS Diagnostic Index
* certain severity of symptoms (at least score of 15 on the International Restless Legs Score (IRLS)
* Have had RLS symptoms for at least 15 nights in the last four weeks.
* < 6 hours of sleep in nights with RLS symptoms
* MADRS (depression rating scale) score of at least 12 (= borderline to depression) at baseline

Exclusion criteria:

* any other sleep disorder that might interfere with the RLS symptoms or sleep (e.g. sleep apnea disorder, narcolepsy)
* Secondary RLS due to diagnosis of renal insufficiency, polyneuropathy, pregnancy (see below), iron deficiency anemia
* Any significant psychiatric disorders (e.g. schizophrenia, bipolar disorder); depression which by judgement of the investigator is caused by RLS, is not an exclusion criterion.
* Current or past suicidality
* medication known to trigger/aggravate/ cause or interfere with RLS symptoms (e.g. most antidepressants, lithium, neuroleptics, opioids, carbidopa, clonidine, antihistamines, anticonvulsants etc.).
* daytime RLS symptoms which require treatment (daytime: 10 a.m. until 6 p.m.).
* concomitant movement disorders (e.g. Parkinson's Disease, dyskinesia, dystonia).
* medical conditions with symptoms which could affect assessments of efficacy (e.g. diabetes, rheumatoid arthritis, fibromyalgia syndrome, cancer etc.).
* Subjects taking any medication known to induce drowsiness or to affect sleep.
* Subjects who are pregnant, lactating or of childbearing potential. Women of childbearing potential must use adequate contraception
* clinically significant or unstable medical conditions (e.g. severe heart disease, severe liver or kidney disease etc.).
* pain syndromes, caused by other disorders than RLS
* excessive caffeine intake
* diastolic blood pressure >110mmHg or <50mmHg or systolic blood pressure >180mmHg or <90mmHg at baseline.
* Withdrawal, introduction, or change in dose of hormone replacement therapy (HRT) or the oral contraceptive pill (OCP) and/or certain drugs which are known to interact with ropinirole (e.g. ciprofloxacin, cimetidine, tobacco, omeprazole).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (37):
- Germany (37):
  - GSK Investigational Site, Ellwangen, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Ostfildern, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Bad Saarow, Brandenburg
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Butzbach, Hesse
  - GSK Investigational Site, Herborn, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Wolfsburg, Lower Saxony
  - GSK Investigational Site, Anklam, Mecklenburg-Vorpommern
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Wismar, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
  - GSK Investigational Site, Jülich, North Rhine-Westphalia
  - GSK Investigational Site, Limburgerhof, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Köthen, Saxony-Anhalt
  - GSK Investigational Site, Oldenburg in Holstein, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Gera, Thuringia
  - GSK Investigational Site, Jena, Thuringia

RESULTS

PARTICIPANT FLOW:
Groups:
- Ropinirole: Subjects who were treated on day 1-2 with 0.25 mg/day of ropinirole and on days 3-7 0.5 mg for 12 weeks if tolerated. After two weeks, dose could be increased weekly by 0.5mg a day up to 4 mg maximum dose.
- Placebo: Subjects who took no investigational product.
Period: Overall Study
Arm/Group | Ropinirole | Placebo
Started | 199 (199 were randomized. Only 198 took investigational product.) | 67
Completed | 145 | 38
Not Completed | 54 | 29
Not completed — Did not meet inclusion criteria | 5 | 3
Not completed — Adverse Event | 34 | 6
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Non-compliance | 1 | 2
Not completed — Lack of Efficacy | 2 | 8
Not completed — Met Exclusion Criteria | 3 | 1
Not completed — Other | 1 | 1
Not completed — Increase of RLS Symptoms | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropinirole | Placebo | Total
Number analyzed (Participants) | 198 | 67 | 265
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (11.4) | 59.5 (11.3) | 58.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 45 | 189.0
  Male | 54 | 22 | 76.0

OUTCOME MEASURES:

1. Primary Outcome: Average Change of the MADRS (Montgomery-Asberg Depression Rating Scale) Total Score From Baseline to Final Visit After 12 Weeks of Treatment
Description: Montgomery-Asberg Depression Rating Scale (MADRS)is a 10 item questionaire preformed during a clinical interview asking broad to detailed questions about symptoms which allows a precise rating of severity of symptoms of the past week. Questions are scored 0-6. Total Score 0-60, the higher the score indicates the most severely depressed patients.
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). The High/Low scores for this population were 32/11.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 171 | 60
Score on a Scale | -10.1 (7.3) | -6.5 (7.6)
Statistical Analysis 1: Comparison: Ropinirole vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -3.6, 95% CI [-5.6 to -1.6] — Mean difference = Ropinirole minus Placebo. Used adjusted change from baseline

2. Secondary Outcome: Average Change of the MADRS (Montgomery-Asberg Depression Rating Scale) Total Score From Baseline to Final Visit After 12 Weeks of Treatment in Participants With Signs of at Least Moderate Depression (MADRS Score: >=18)
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). Sub-population with MADRS scores>=18: Ropinirole 91 and Placebo 29. The high/Low scores for the mITT population were 32/11.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 91 | 29
Score on a Scale | -12.5 (8.0) | -8.8 (9.2)

3. Secondary Outcome: Average Change of the HAM-D (Hamilton Depression Rating Scale, 17-item-Version) Total Score From Baseline to Final Visit After 12 Weeks of Treatment
Description: The Hamilton Rating Scale for Depression contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAMD score range from 0 (not ill) to 54 (severely ill).
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). The High/Low HAM-D scores for this population were 27/5.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 166 | 55
Score on a Scale | -8.2 (5.5) | -5.5 (6.4)

4. Secondary Outcome: Average Change of the HAM-D Total Score From Baseline to Final Visit After 12 Weeks of Treatment in Participants With Signs of an at Least Moderate Depression (HAM-D Score >= 15) at Baseline
Description: The Hamilton Rating Scale for Depression contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAMD score range from 0 (not ill) to 54(severely ill).
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). Sub-population with HAM-D scores>=15: Ropinirole 93 and Placebo 33
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 93 | 33
Score on a Scale | -9.6 (5.9) | -7.2 (6.6)

5. Secondary Outcome: Average Change of the Beck Depression Inventory (BDI) Total Score From Baseline to Final Visit After 12 Weeks of Treatment
Description: Becks Depression Inventory (BDI) is a 21 item self inventory evaluating symptoms of depression, cognition, and physical symptoms of fatigue, weight loss, and lack of interest in sex. The Higher the score represents most severely depressed participants. Score range for each items is 0-3 and Total score 0-63.
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). High/Low BDI scores for this population were 46/2.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 169 | 60
Score on a Scale | -8.6 (7.0) | -6.5 (7.8)

6. Secondary Outcome: Average Change of the Beck Depression Inventory (BDI) Total Score From Baseline to Final Visit After 12 Weeks of Treatment in Participants With Signs of an at Least Mild-moderate Depression (BDI >= 21) at Baseline
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). Sub-population with BDI scores>=21: Ropinirole 75 and Placebo 28. High/Low BDI scores for this population were 46/2.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 75 | 28
Score on a Scale | -10.9 (7.9) | -9.9 (9.0)

7. Secondary Outcome: Percentage of Participants With at Least Moderate Depression (MADRS Score >= 18) at Baseline and in Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at week 12).
Measure: Number; unit: Percentage of Participants
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 171 | 60
Percentage of Participants | 11.7 | 23.3

8. Secondary Outcome: Percentage of Participants With at Least Moderate Depression (HAM-D >= 15) at Baseline and in Week 12
Description: as for outcome 3
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). Sub-population with HAM-D scores>=15.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 168 | 56
Percentage of Participants | 10.7 | 26.8

9. Secondary Outcome: Percentage of Participants ("Responder") With a Decrease of MADRS Total Score of at Least 6 Points After 12 Weeks Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5).
Measure: Number; unit: Percentage of Participants
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 171 | 60
Percentage of Participants | 74.9 | 48.3

10. Secondary Outcome: Percentage of Participants ("Responder") With a Decrease of MADRS Total Score of at Least 6 Points After 12 Weeks Compared to Baseline in Subjects With Signs of at Least Moderate Depression at Baseline (MADRS Score >= 18)
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). Sub-population with MADRS scores>=18: Ropinirole 91 and Placebo 29
Measure: Number; unit: Percentage of Participants
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 91 | 29
Percentage of Participants | 80.2 | 58.6

11. Secondary Outcome: Change in Average MADRS Score From Baseline to Final Visit (Week 12) in Participants With Major Depressive Episodes (Diagnosed by MINI Interview Modules A, B and C / DSM Criteria)
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). Sub-population diagnosed by MINI interview with Major Depressive Episodes: Ropinirole 93 and Placebo 34
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 93 | 34
Score on a Scale | -11.6 (7.7) | -7.6 (8.1)

12. Secondary Outcome: Change in Average HAM-D Score From Baseline to Final Visit (Week 12) in Participants With Major Depressive Episodes (Diagnosed by MINI Interview Modules A, B and C / DSM Criteria)
Description: as for outcome 3
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). Sub-population diagnosed by MINI interview with Major Depressive Episodes: Ropinirole 90 and Placebo 31.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 90 | 31
Score on a Scale | -9.2 (5.6) | -6.5 (7.0)

13. Secondary Outcome: Change in Average BDI Score From Baseline to Final Visit (Week 12) in Participants With Major Depressive Episodes (Diagnosed by MINI Interview Modules A, B and C / DSM Criteria)
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: Modified Intent to Treat (mITT): All treated patients with MADRS score at baseline and post baseline (i.e., at visit 4 and/or 5). Sub-population diagnosed by MINI interview with Major Depressive Episodes: Ropinirole 91 and Placebo 34. High/Low BDI scores for this population were 46/2.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 91 | 34
Score on a Scale | -10.4 (6.8) | -7.2 (8.2)

14. Secondary Outcome: Change in Average International Restless Legs Scale for Severity (IRLS) Scores in All Participants From Baseline to After 1, 4, and 12 Weeks
Description: International Restless Legs Scale for Severity (IRLS)is a series of 10 questions which rate severity from 0-4 points for various questions and total score ranks: Very severe=31-40 points, Severe=21-30 points, Moderate=11-20 points, and Mild=1-10 points, None=0 points
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: Intent to Treat (ITT): All patients of the safety population with any psychometric data at baseline (within a single questionnaire)
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 171 | 60
Score on a Scale
  Change from Baseline after 1 Week | -7.7 (8.0) | -4.1 (5.4)
  Change from Baseline after 4 Weeks | -14.0 (9.2) | -8.6 (8.5)
  Change from Baseline after 12 Weeks | -14.6 (9.2) | -10.2 (10.6)

15. Secondary Outcome: Percentage of Participants With a Decrease of International Restless Legs Scale (IRLS) Scores of at Least 6 Points After 1, 4 and 12 Weeks
Description: as for outcome 14
Time Frame: Week 1, Week 4, Week 12
Population: as for outcome 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 171 | 60
Percentage of Participants
  1 Week | 52.6 | 28.3
  4 Weeks | 80.7 | 58.3
  12 Weeks | 84.8 | 61.7

16. Secondary Outcome: Percentage of Participants With "Much Improved" or "Very Much Improved" on the Clinical Global Impression-Global Improvement Scale After 1, 4 and 12 Weeks
Description: The CGI-I assesses the investigator's impression of the patient's current illness. The time span is the week before the rating and the score range: 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5- minimally worse, 6-much worse, to 7-very much worse.
Time Frame: Week 1, Week 4, Week 12
Population: as for outcome 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 171 | 60
Percentage of Participants
  Week 1 | 35.1 | 15.0
  Week 4 | 66.7 | 40.0
  Week 12 | 64.3 | 46.7

17. Secondary Outcome: Change From Average Baseline Score of Subscale of "Somnolence" in the Medical Outcomes Study Sleep Scale (MOS-SS) to Final Visit After 12 Weeks
Description: Medical Outcome Study Sleep Scale (MOS-SS)-is a 12 item questionaire assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache. 10 question score from 1-6, 1 question scores 1-5 and 1 question asks average number of hours sleep each night.
Time Frame: Baseline and after Week 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 171 | 59
Score on a Scale | -12.5 (19.4) | -10.2 (19.9)

18. Secondary Outcome: Change From Average Baseline Scores of Subscale "Sleep Disturbance" of the Medical Outcomes Study Sleep Scale (MOS-SS) to Final Visit After 12 Weeks
Description: as for outcome 17
Time Frame: Baseline and after Week 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 167 | 59
Score on a Scale | -30.5 (24.5) | -15.8 (27.6)

19. Secondary Outcome: Change From Average Baseline Scores of Subscale "Sleep Adequacy" of the Medical Outcomes Study Sleep Scale (MOS-SS)to Final Visit After 12 Weeks
Description: as for outcome 17
Time Frame: Baseline and after Week 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 170 | 59
Score on a Scale | 34.0 (30.6) | 15.6 (36.2)

20. Secondary Outcome: Change From Average Baseline Scores of Subscale "Sleep Quantity" (Hours) of the Medical Outcomes Study Sleep Scale (MOS-SS) to Final Visit After 12 Weeks
Time Frame: Baseline and after Week 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ropinirole | Placebo
Number analyzed (Participants) | 170 | 59
Score on a Scale | 1.3 (1.3) | 0.5 (1.4)

ADVERSE EVENTS:
Arm/Group | Ropinirole | Placebo
Serious Adverse Events (participants affected / at risk) | 4 | 0
Other Adverse Events (participants affected / at risk) | 134 | 20
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Ropinirole | Placebo
Back Pain (Respiratory, thoracic and mediastinal disorders) | 1/197 | 0/67
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1/197 | 0/67
Nausea (Gastrointestinal disorders) | 1/197 | 0/67
Vomiting (Gastrointestinal disorders) | 1/197 | 0/67
Bronchitis (Infections and infestations) | 1/197 (1) | 0/67 (0)
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 1/197 (1) | 0/67 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Ropinirole | Placebo
Nausea (Gastrointestinal disorders) | 64/197 | 5/67
Vomiting (Gastrointestinal disorders) | 14/197 | 0/67
Fatigue (General disorders) | 25/197 | 4/67
Dizziness (Nervous system disorders) | 17/197 | 2/67
Headache (Nervous system disorders) | 39/197 | 9/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.